CLINICAL TRIAL: NCT06882889
Title: A Non-Inferiority, Single-Blind, Randomized Controlled Trial Comparing the Efficacy of Domestic Versus Imported Hearing Aids in Patients With Moderate to Severe and Severe Age-Related Hearing Loss
Brief Title: Comparing the Efficacy of Domestic Versus Imported Hearing Aids in ARHL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2024-761-02
Record Dates: First submitted 2025-02-11; First posted 2025-03-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Age-related Hearing Loss; Hearing Loss, Sensorineural
Keywords: Age-related hearing loss; Hearing Aids; Randomized Controlled Trial
MeSH Terms: conditions — Presbycusis; Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: The experimental group will use domestic hearing aids, and the control group will use imported hearing aids.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group will use domestic hearing aids.
  Interventions: Device: Domestic hearing aids
- The control group (Active Comparator): The control group will use imported hearing aids.
  Interventions: Device: Imported hearing aids

INTERVENTIONS:
Device: Domestic hearing aids — The domestic hearing aids used in this study are from the Bigsound brand. Using domestic hearing aids for intervention, one first evaluates the patient's hearing condition through pure-tone audiometry. Subsequently, by thoroughly understanding the patient's hearing needs, lifestyle, and other relevant factors, the most suitable type and functions of hearing aids are selected to best meet the individual's specific situation.
  Arms: The experimental group
Device: Imported hearing aids — The imported hearing aids used in this study are from the Phonak brand. Using imported hearing aids for intervention, one first evaluates the patient's hearing condition through pure-tone audiometry. Then, by thoroughly understanding the patient's hearing needs, lifestyle, and other relevant factors, the most suitable type and functions of hearing aids are selected to best meet the individual's specific situation.
  Arms: The control group

SUMMARY:
This study compares the hearing improvement effects of domestic hearing aids and imported hearing aids in 80 patients with moderate to severe and severe age-related hearing loss. Patients will be randomly assigned to either the experimental group (domestic hearing aids) or the control group (imported hearing aids) and will undergo a 30-minute trial. Pure Tone Average (PTA) and Speech Recognition Threshold (SRT) will be measured both before and after the trial. The improvements in PTA and SRT will be calculated.The market prices of the hearing aids and the degree of hearing improvement in decibels will be recorded. These data will be used to conduct a comprehensive cost-effectiveness analysis. After the trial, the International Outcome Inventory for Hearing Aids (IOI-HA) and the Abbreviated Profile of Hearing Aid Benefit (APHAB) will be used to assess the benefits of the hearing aids.

DETAILED DESCRIPTION:
This study aims to conduct a non-inferiority, single-blind, randomized controlled trial to compare the hearing improvement effects of domestic hearing aids versus imported hearing aids in patients with moderate to severe and severe age-related hearing loss.

A total of 80 patients meeting the inclusion and exclusion criteria will be randomly assigned to either the experimental group (domestic hearing aids) or the control group (imported hearing aids).

The domestic hearing aids used in this study are from the Bigsound brand and include behind-the-ear (BTE), neck-worn, and in-the-ear (ITE) styles. All of these hearing aids are rechargeable.The imported hearing aids used in this study are from the Phonak brand and include behind-the-ear (BTE), neck-worn, and in-the-ear (ITE) styles.

Each group will undergo a 30-minute trial with their respective hearing aids. Pure Tone Average (PTA) and Speech Recognition Threshold (SRT) before and after the 30-minute trial will be collected, and the improvements in PTA and SRT will be calculated.The market price of the hearing aids and the degree of hearing improvement in decibels for each patient will be recorded, and a comprehensive cost-effectiveness analysis will be performed. Additionally, after the 30-minute trial, the International Outcome Inventory for Hearing Aids (IOI-HA) and the Abbreviated Profile of Hearing Aid Benefit (APHAB) will be used to assess the benefits of the hearing aids.

Statistical analyses will be conducted to determine whether the domestic hearing aids are non-inferior to the imported hearing aids in terms of hearing and speech improvement. The analysis will also evaluate patient satisfaction, performance in different listening environments, and adaptation to the hearing aids for both the domestic hearing aids and imported hearing aids.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years and ≤ 85 years;
2. Diagnosed with age-related hearing Loss, which is characterized by bilateral, symmetrical, and gradually progressive hearing loss primarily affecting high frequencies, along with a decline in speech recognition ability, as referenced in the "Expert Consensus on Diagnosis and Intervention of Age-Related Hearing Loss" (2019 edition);
3. Age-related hearing Loss is of moderate to severe or severe sensorineural hearing loss, with moderate to severe defined as 50 to <65 dB HL, and severe defined as 65 to <80 dB HL;
4. Chinese nationality, able to complete all assessments in the Chinese language;
5. Right-handed;
6. No significant neurological diseases, severe systemic diseases, family history of genetic disorders, or major psychiatric conditions;

Exclusion Criteria:

1. Exclusion of noise-induced hearing loss, hereditary hearing loss, drug-induced hearing loss, etc.;
2. Inability to use hearing aids ;
3. Presence of dementia, Parkinson's disease, or other neurodegenerative diseases that may affect study compliance;
4. History of cerebrovascular accidents, stroke, epilepsy, or other central nervous system disorders;
5. Other conditions deemed by the investigator to be exclusionary.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Pure Tone Average (ΔPTA) | The initial assessment will be conducted prior to the use of the hearing aid, and the follow-up assessment will be performed 0.5 hours after the hearing aid is used.
  Improvement in Pure Tone Average (ΔPTA):
  The improvement in Pure Tone Average (ΔPTA) will be assessed by measuring the average of the lowest sound intensities detectable at 0.5 kHz, 1 kHz, 2 kHz, and 4 kHz in the better ear of patients with moderate to severe and severe age-related hearing loss both before and after hearing aid fitting, using pure tone audiometry and sound field audiometry. These measurements will be recorded as pre-fitting PTA and post-fitting PTA.
  Improvement in Pure Tone Average (ΔPTA) = post-fitting PTA - pre-fitting PTA

SECONDARY OUTCOMES:
Improvement in Speech Recognition Threshold (ΔSRT) | The initial assessment will be conducted prior to the use of the hearing aid, and the follow-up assessment will be performed 0.5 hours after the hearing aid is used.
  Improvement in Speech Recognition Threshold (ΔSRT):
  The improvement in Speech Recognition Threshold (ΔSRT) will be assessed by measuring the lowest sound intensity at which 50% of spondee words are correctly identified by patients with moderate to severe and severe age-related hearing loss , both before and after hearing aid fitting. This will be done using speech audiometry and sound field speech audiometry. The measurements will be recorded as pre-fitting SRT and post-fitting SRT.
  Improvement in Speech Recognition Threshold (ΔSRT)= post-fitting SRT - pre-fitting SRT
International Outcome Inventory for Hearing Aids (IOI-HA) | The assessment will be conducted only after the patient has used the hearing aid for 0.5 hours.
  The International Outcome Inventory for Hearing Aids (IOI-HA) scale will be used to evaluate the usage experience and satisfaction of patients with moderate to severe and severe age-related hearing loss after wearing domestic hearing aids and imported hearing aids for 30 minutes.
Abbreviated Profile of Hearing Aid Benefit (APHAB) | The assessment will be conducted only after the patient has used the hearing aid for 0.5 hours.
  Abbreviated Profile of Hearing Aid Benefit (APHAB) :
  The Abbreviated Profile of Hearing Aid Benefit (APHAB) scale will be used to evaluate the hearing performance of patients with moderate to severe and severe age-related hearing loss in different listening situations after wearing domestic hearing aids and imported hearing aids for 0.5 hours. This assessment aims to understand the effectiveness of the hearing aids in various listening environments and the patients' adaptation to the hearing aids.
Cost-Effectiveness Analysis (CEA): | The assessment will be conducted only after the patient has used the hearing aid for 0.5 hours.
  Cost-Effectiveness Analysis (CEA) will be used to evaluate the estimated costs of domestic hearing aids and imported hearing aids. The degree of hearing loss in decibels (dB) for patients with moderate to severe and severe age-related hearing loss will be recorded. The cost-effectiveness ratio will be calculated by dividing the total costs by the number of dB of hearing improvement. The measurement will be in Chinese Yuan (CNY) per dB.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Haidi, PhD, Study Chair — SunYatSunU2H
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No